CLINICAL TRIAL: NCT07327840
Title: A Double-blind, Randomized, Placebo-controlled Phase 2 Study to Evaluate Efficacy and Safety of Kylo-11 in Participants With Atherosclerotic Cardiovascular Disease and Elevated Lipoprotein(a)
Brief Title: Phase 2 Study of Kylo-11 in ASCVD Patients With Elevated Lp(a)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kylonova (Xiamen) Biopharma co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kylo-11-II-C01
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Lipoprotein Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Kylo-11 dose 1 or matched placebo will be administered subcutaneously
  Interventions: Drug: Kylo-11 or matched placebo
- Cohort 2 (Experimental): Kylo-11 dose 2 or matched placebo will be administered subcutaneously
  Interventions: Drug: Kylo-11 or matched placebo
- Cohort 3 (Experimental): Kylo-11 dose 3 or matched placebo will be administered subcutaneously
  Interventions: Drug: Kylo-11 or matched placebo

INTERVENTIONS:
Drug: Kylo-11 or matched placebo — Administered subcutaneously

SUMMARY:
This is a phase 2, double-blind, randomized, placebo-controlled, multi-center, dose-finding study to evaluate the efficacy and safety of Kylo-11 administered subcutaneously compared to placebo in participants with ASCVD and elevated Lp(a).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years
* Clinical diagnosis of atherosclerotic cardiovascular disease with elevated Lp(a)
* Other inclusion criteria applied per protocol.

Exclusion Criteria:

* Have moderate to severe heart failure (New York Heart Association [NYHA] Functional Classification III or IV during Screening) or last known left ventricular ejection fraction <30%
* Have uncontrolled hypertension (systolic blood pressure [SBP] ≥160 mmHg or diastolic blood pressure [DBP] ≥100 mmHg)
* Have uncontrolled cardiac arrhythmia defined as recurrent and highly symptomatic ventricular tachycardia, atrial fibrillation with rapid ventricular response, or supraventricular tachycardia that are not controlled by medications, in the past 3 months prior to randomization
* Have had any malignancy within 5 years prior to randomization (except for non-melanoma skin cancers, cervical in-situ carcinoma, breast ductal carcinoma in situ, or stage 1 prostate carcinoma that has been successfully treated)
* Other exclusion criteria applied per protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in time-averaged Lp(a) over Weeks 8~26 | Baseline, Weeks 8~26
  A MMRM including terms of treatment arm, stratification factors, scheduled visit and the interaction of treatment arm with scheduled visit will be used to estimate the percent change from baseline in time-averaged Lp(a) over Weeks 8~26. The least squares means (LS means) by treatment arm and the treatment difference (Kylo-11 - placebo) based on the model will be summarized.

SECONDARY OUTCOMES:
Percent change from baseline in time-averaged Lp(a) over Weeks 38~52 | Baseline, Weeks 38~52
  A MMRM including terms of treatment arm, stratification factors, scheduled visit and the interaction of treatment arm with scheduled visit will be used to estimate the percent change from baseline in time-averaged Lp(a) over Weeks 8~26. The least squares means (LS means) by treatment arm and the treatment difference (Kylo-11 - placebo) based on the model will be summarized.
Proportion of participants achieving Lp(a) <125 nmol/L and <75 nmol/L at Week 26 and Week 52 | Week 26 and Week 52
  For proportion of participants achieving Lp(a) <125 nmol/L and <75 nmol/L at Week 26 and Week 52, the number of responders in both the Kylo-11 arm and the placebo arm will be calculated separately.

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Baotou Medical College, Baotou
  - Beijing Anzhen Hospital, Beijing
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing
  - Chongqing University Three Gorges Hospital, Chongqing
  - The First Affiliated Hospital of Dali University, Dali
  - Daqingshi People's Hospital, Daqing
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - The First Affiliated Hospital of University of South China, Hengyang
  - Central Hospital Affiliated to Shandong First Medical University, Jinan
  - Luoyang Third People's Hospital, Luoyang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Nanchang People's Hospital, Nanchang
  - Nanyang Medical College First Affiliated Hospital, Nanyang
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Hainan Third People's Hospital, Sanya
  - Tongji Medical College of Hust Tongji Hospital, Wuhan
  - Shaanxi Provincial People's Hospital, Xi'an
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen
  - Yuncheng Central Hospital of Shanxi Province, Yuncheng
  - Zibo Central Hospital, Zibo

IPD SHARING:
Plan to Share IPD: No